CLINICAL TRIAL: NCT05278130
Title: Serial Screening and Treatment of Bacterial Vaginosis in Pregnancy to Prevent Preterm Delivery: A Randomized Control Trial
Brief Title: Serial Screening and Treatment of Bacterial Vaginosis Trial
Acronym: SECRETIVA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated/no study participants were ever enrolled.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5220115
Record Dates: First submitted 2022-01-21; First posted 2022-03-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Bacterial Vaginosis; Preterm Delivery
Keywords: Bacterial Vaginosis; Vaginoses, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): The intervention-arm will have a pelvic exam performed with vaginal swab collection at their initial obstetric visit (standard of care). The women undergoing the intervention will then subsequently undergo additional vaginal swab collections in 2 week intervals starting at 16 weeks gestational age until 34 weeks gestational age. Subjects will be informed of the results of the vaginal swab. If positive for an infection, subjects will be provided with the appropriate treatment in pregnancy.
  Interventions: Other: Additional vaginal swabs
- Control Arm (No Intervention): The control arm will undergo the standard of care with vaginal swab collection at their initial obstetric visit. The control arm will not undergo additional vaginal swab collections unless otherwise indicated under standard of care (further testing for bacterial vaginosis is completed in women who describe symptoms with the diagnosis or present for preterm contractions and/or pelvic cramping). There will be no placebo for the control group.

INTERVENTIONS:
Other: Additional vaginal swabs — Every 2 weeks from 16 weeks gestational age to 34 weeks gestational age
  Arms: Intervention Arm

SUMMARY:
The purpose of this investigator-initiated randomized control trial is to determine if bacterial vaginosis infection increases the likelihood of preterm delivery in women with history of preterm delivery. Subjects will be randomized in a two-arm study to undergo predetermined intervals of testing for bacterial vaginosis or control.

DETAILED DESCRIPTION:
Preterm delivery affects 10% of all pregnancies in the United States. This risk is further increased in pregnant women with a history of preterm delivery. There are multiple etiology contributing of preterm labor. Of these, the presence of inflammation and infection have been a well-established cause. Bacterial vaginosis (BV), a common vaginal infection in pregnancy, may often be asymptomatic. Studies demonstrate a strong association between BV and preterm labor. Therefore it is recommended that women at high risk for preterm delivery are treated for this infection irregardless of symptoms. In this study the investigators hypothesize that increased testing for bacterial vaginosis, with subsequent timely treatment, may decrease the risk of preterm delivery in patients who are at high risk. The investigators suspect that the increase in monitoring will help diagnose asymptomatic bacterial vaginosis infections allowing for prompt treatment and avoidance of preterm labor.

Subjects will be randomized in a two-arm study to undergo predetermined intervals of testing for bacterial vaginosis or control. No experimental drugs or devices will be used.

* The intervention-arm will have a pelvic exam performed with vaginal swab collection at their initial obstetric visit. The women undergoing the intervention will then subsequently undergo additional vaginal swab collections in 2 week intervals starting at 16 weeks gestational age until 34 weeks gestational age.
* The control arm will undergo the standard of care. There will be no placebo for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age greater than or equal to 18 years old
* Pregnancy at less than 32 weeks gestational age at initial obstetric visit with Loma Linda Maternal Fetal Medicine (MFM) Clinic
* History of at least one prior preterm delivery >16 and <37 weeks not due to iatrogenic indications, or short cervical length <2.5cm
* Willing to receive prenatal standard of care and comply with treatment plan and other study procedures at Loma Linda

Exclusion Criteria:

* Patients not deemed to be high risk for preterm delivery
* Patient with cervical dilation ≥1cm on initial exam or with protruding membranes
* Current pregnancy is multigestation
* Medical indications for iatrogenic preterm delivery during this pregnancy (e.g. preeclampsia with severe features)
* Desires termination during this pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with premature delivery (before 37 weeks gestation) | At delivery

OTHER OUTCOMES:
Length of hospital stay of mothers | Number of hours between time of admission to time of discharge, up to 4 weeks from time of admission
  The length of hospital stay for mothers will be measured in hours from the time of admission to labor and delivery unit to the time of discharge from the post-partum unit.
Length of hospital stay of neonates | Number of hours between time of admission (birth) to time of discharge, up to 1 year from time of admission (birth)
  The length of hospital stay for neonates will be measured in hours from the time of admission (birth) to discharge from the postpartum unit or neonatal intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No